CLINICAL TRIAL: NCT00003516
Title: Phase II Study of Antineoplaston A10 and AS2-1 Capsules In Patients With Incurable, Stage C or D Adenocarcinoma of the Prostate
Brief Title: Antineoplaston Therapy in Treating Patients With Stage III or Stage IV Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066559; BC-PR-5 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: Stage III or Stage IV Prostate Cancer Stage III; Stage III or Stage IV Prostate Cancer Stage IV
MeSH Terms: conditions — Prostatic Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplastons (Experimental): Antineoplaston therapy (Atengenal + Astugenal) capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity. absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Antineoplaston therapy (Atengenal + Astugenal) capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity. absence of disease progression or unacceptable toxicity.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Stage III or Stage IV Prostate Cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage III or Stage IV Prostate Cancer.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage III or Stage IV Prostate Cancer.

DETAILED DESCRIPTION:
Stage III or Stage IV Prostate Cancers receive Antineoplaston A10 and AS2-1 capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage III or Stage IV Prostate Cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage III or Stage IV Prostate Cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 4 months for 2 years, every 6 months for 2 years, and then annually for 2 years thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage III or IV adenocarcinoma of the prostate not potentially curable by surgery or radiotherapy
* Measurable tumors or tumor markers
* No response to antiandrogen withdrawal

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT no greater than 2 times normal
* No hepatic failure

Renal:

* BUN less than 60 mg/dL
* Creatinine no greater than 2.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* Blood ammonia normal
* No chronic renal failure

Cardiovascular:

* No severe heart disease

Pulmonary:

* No severe lung disease

Other:

* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infection or fever
* No other concurrent serious disease
* No other prior or concurrent malignancy within the past 2 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy and recovered
* Prior corticosteroids for at least 2 months allowed, but must be on stable or decreasing dose during study participation

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery and recovered

Other:

* At least 4 weeks since prior experimental clinical trial
* No other concurrent therapy for metastatic disease

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1996-03-27 (Actual); Primary Completion 2004-03-18 (Actual); Study Completion 2004-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com